CLINICAL TRIAL: NCT03424109
Title: Primary Palliative Care for Emergency Medicine (PRIM-ER)
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-00607; 5UH3AT009844 (NIH); NCT03424096 (obsolete NCT alias)
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Emergencies
Keywords: Emergency Department; Palliative Care
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Beneficiaries with a one-year mortality of at least 30%: The patient cohort will be extracted via the Centers for Medicare and Medicaid Services (CMS) Research Data Assistance Center (ResDAC) using a two-step process to maximize diversity, and minimize intentional or unintentional exclusions based on risk, age, health literacy, demographics, or expected adherence.
  Interventions: Behavioral: healthcare service utilization in the six months following the ED visit

INTERVENTIONS:
Behavioral: healthcare service utilization in the six months following the ED visit — The analysis of the effect of PRIM-ER on ED disposition using a generalized linear binomial model with random site level effects.

SUMMARY:
This proposal builds upon the evaluation of Primary Palliative Care Education, Training, and Technical Support for Emergency Medicine (PRIM-ER) implemented in a cluster-randomized, stepped wedge design in 33 Emergency Departments (EDs).

ELIGIBILITY:
Inclusion Criteria:

* Patients must demonstrate one-year mortality of at least 30 percent (score > 6) according to the Gagne Index, a validated instrument used to measure all cause one-year mortality in community-dwelling older adults, calculated based on their prior 12 months before the index ED visit of Medicare claims.

Exclusion Criteria:

* ED patients transferred from a nursing home on the index ED visit will be excluded since prediction of mortality and disposition of such patients differs from community-dwelling adults.
* Patients currently receiving hospice at the time of the index ED visit will also be excluded since they have already received services.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Eligible patients will include ED patients 66 years or older with serious, life-limiting illness who visited any of our EDs during the implementation of PRIM-ER.
Sampling Method: Non-Probability Sample
Enrollment: 98922 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith S Goldfeld, DrPH, MS, MPA, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share all policies, practices, materials, and tools to facilitate collaboration, reuse, and replication, including clinical workflows, design specifications for our clinical decision support and learning management system, code sets for extraction, and definition of data from Medicare administrative claims. PI will comply with the ResDAC VRDC rules regarding the sharing and reporting of data in aggregate form only. A final dataset will not be available for collaboration, reuse, and replication of the findings because of our decision to use the ResDAC VRDC.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Grudzen CR, Siman N, Cuthel AM, Adeyemi O, Yamarik RL, Goldfeld KS; PRIM-ER Investigators; Abella BS, Bellolio F, Bourenane S, Brody AA, Cameron-Comasco L, Chodosh J, Cooper JJ, Deutsch AL, Elie MC, Elsayem A, Fernandez R, Fleischer-Black J, Gang M, Genes N, Goett R, Heaton H, Hill J, Horwitz L, Isaacs E, Jubanyik K, Lamba S, Lawrence K, Lin M, Loprinzi-Brauer C, Madsen T, Miller J, Modrek A, Otero R, Ouchi K, Richardson C, Richardson LD, Ryan M, Schoenfeld E, Shaw M, Shreves A, Southerland LT, Tan A, Uspal J, Venkat A, Walker L, Wittman I, Zimny E. Palliative Care Initiated in the Emergency Department: A Cluster Randomized Clinical Trial. JAMA. 2025 Feb 18;333(7):599-608. doi: 10.1001/jama.2024.23696. PMID 39813042
- [Derived] Adeyemi O, Ginsburg AD, Kaur R, Cuthel AM, Zhao N, Siman N, Goldfeld KS, Emlet LL, DiMaggio C, Yamarik RL, Bouillon-Minois JB, Chodosh J, Grudzen CR; PRIM-E. R. Investigators. Serious illness communication skills training for emergency physicians and advanced practice providers: a multi-method assessment of the reach and effectiveness of the intervention. BMC Palliat Care. 2024 Feb 21;23(1):48. doi: 10.1186/s12904-024-01349-y. PMID 38378532
- [Derived] Adeyemi OJ, Siman N, Goldfeld KS, Cuthel AM, Bouillon-Minois JB, Grudzen CR. Emergency Providers' Knowledge and Attitudes Toward Hospice and Palliative Care: A Cross-Sectional Analysis Across 35 Emergency Departments in the United States. J Palliat Med. 2023 Sep;26(9):1252-1260. doi: 10.1089/jpm.2022.0545. Epub 2023 Jun 1. PMID 37262130
- [Derived] Adeyemi O, Ginsburg AD, Kaur R, Cuthel A, Zhao N, Siman N, Goldfeld K, Emlet LL, DiMaggio C, Yamarik R, Bouillon-Minois JB, Chodosh J, Grudzen CR; PRIM-ER Investigators. Serious Illness Communication Skills Training for Emergency Physicians and Advanced Practice Providers: A Multi-Method Assessment of the Reach and Effectiveness of the Intervention. Res Sq [Preprint]. 2023 Feb 21:rs.3.rs-2561749. doi: 10.21203/rs.3.rs-2561749/v1. PMID 36865121
- [Derived] Chung FR, Turecamo S, Cuthel AM, Grudzen CR; PRIM-ER Investigators. Effectiveness and Reach of the Primary Palliative Care for Emergency Medicine (PRIM-ER) Pilot Study: a Qualitative Analysis. J Gen Intern Med. 2021 Feb;36(2):296-304. doi: 10.1007/s11606-020-06302-2. Epub 2020 Oct 27. PMID 33111240
- [Derived] Tan A, Durbin M, Chung FR, Rubin AL, Cuthel AM, McQuilkin JA, Modrek AS, Jamin C, Gavin N, Mann D, Swartz JL, Austrian JS, Testa PA, Hill JD, Grudzen CR; Group Authorship: Corita R. Grudzen on behalf of the PRIM-ER Clinical Informatics Advisory Board. Design and implementation of a clinical decision support tool for primary palliative Care for Emergency Medicine (PRIM-ER). BMC Med Inform Decis Mak. 2020 Jan 28;20(1):13. doi: 10.1186/s12911-020-1021-7. PMID 31992301
- [Derived] Grudzen CR, Brody AA, Chung FR, Cuthel AM, Mann D, McQuilkin JA, Rubin AL, Swartz J, Tan A, Goldfeld KS; PRIM-ER Investigators. Primary Palliative Care for Emergency Medicine (PRIM-ER): Protocol for a Pragmatic, Cluster-Randomised, Stepped Wedge Design to Test the Effectiveness of Primary Palliative Care Education, Training and Technical Support for Emergency Medicine. BMJ Open. 2019 Jul 27;9(7):e030099. doi: 10.1136/bmjopen-2019-030099. PMID 31352424

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an **observational** cluster-randomized **quality improvement (QI) initiative**. Randomization of patients occurred at the ED level; EDs (and subsequent visiting patients) were assigned to either "Control" (i.e., no intervention) or "PRIM-ER" (intervention). Medicare claims of the beneficiaries (visiting patients) from index visit and the six months following the index visit were analyzed to assess outcomes. Participant flow data is not analyzed by sequence but rather by arm/condition.
Units Other Than Participants: Emergency Departments
Groups:
- Control for Six Months, Then PRIM-ER: Care as usual for six months - participants did not cross over.
  At six months, intervention comprising primary palliative care education, training, and technical support for emergency medicine (PRIM-ER) implemented at participating emergency departments.
Period: Control Period
Arm/Group | Control for Six Months, Then PRIM-ER
Started | 50458; 33 Emergency Departments
Completed | 50458; 33 Emergency Departments
Not Completed | 0; 0 Emergency Departments
Period: PRIM-ER Intervention Period
Arm/Group | Control for Six Months, Then PRIM-ER
Started | 48464; 33 Emergency Departments
Completed | 48464; 33 Emergency Departments
Not Completed | 0; 0 Emergency Departments

BASELINE CHARACTERISTICS:
Groups:
- Control: Care as usual.
  -ER).
- PRIM-ER: Intervention comprising primary palliative care education, training, and technical support for emergency medicine (PRIM-ER).
- Total: Total of all reporting groups
Arm/Group | Control | PRIM-ER | Total
Number analyzed (Participants) | 50458 | 48464 | 98922
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.2 (8.5) | 77.7 (8.3) | 78 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25137 | 23904 | 49041
  Male | 25321 | 24560 | 49881
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 735 | 727 | 1462
  Not Hispanic or Latino | 49723 | 47737 | 97460
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 93 | 60 | 153
  Asian | 1555 | 1233 | 2788
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6341 | 7006 | 13347
  White | 39642 | 37308 | 76950
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2827 | 2857 | 5684
Region of Enrollment [Number; unit: participants]
  United States | 50458 | 48464 | 98922

OUTCOME MEASURES:

1. Primary Outcome: Acute Care Admission
Description: Proportion of eligible patients whose disposition is to an acute care setting (inpatient, non-palliative service).
Time Frame: Index Visit
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Emergency Departments (EDs)
Groups:
- Control: Patients who received care as usual.
- PRIM-ER: Patients who received PRIM-ER.
Arm/Group | Control | PRIM-ER
Number analyzed (Participants) | 50458 | 48464
Number analyzed (Emergency Departments (EDs)) | 33 | 33
Proportion of participants | 0.644 | 0.613

2. Secondary Outcome: Proportion of Patients With Emergency Department (ED) Revisits
Description: Measured as the proportion of patients with at least one ED revisit in the six months following the index ED visit (Count)
Time Frame: Up to Month 6
Measure: Number; unit: Proportion of Patients
Units Other Than Participants: Emergency Departments (EDs)
Arm/Group | Control | PRIM-ER
Number analyzed (Participants) | 50458 | 48464
Number analyzed (Emergency Departments (EDs)) | 33 | 33
Proportion of Patients | 0.6 | 0.6

3. Secondary Outcome: Inpatient Days
Description: Measured as the proportion of patients who had at least one inpatient stay in the six months following the index ED visit (Count).
Time Frame: Up to Month 6
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Emergency Departments (EDs)
Arm/Group | Control | PRIM-ER
Number analyzed (Participants) | 50458 | 48464
Number analyzed (Emergency Departments (EDs)) | 33 | 33
Proportion of participants | 0.410 | 0.366

4. Secondary Outcome: Home Health Use
Description: Proportion of patients with any home health use in the six months following the index ED visit (Yes/No)
Time Frame: Up to Month 6
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Emergency Departments (EDs)
Arm/Group | Control | PRIM-ER
Number analyzed (Participants) | 50458 | 48464
Number analyzed (Emergency Departments (EDs)) | 33 | 33
Proportion of participants | 0.420 | 0.381

5. Secondary Outcome: Hospice Use
Description: Proportion of patients with any hospice use in the six months following the index ED visit (Yes/No).
Time Frame: Up to Month 6
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Emergency Departments (EDs)
Arm/Group | Control | PRIM-ER
Number analyzed (Participants) | 50458 | 48464
Number analyzed (Emergency Departments (EDs)) | 33 | 33
Proportion of participants | 0.177 | 0.172

6. Secondary Outcome: Proportion of Patients Who Died at Month 6 Post-Index Visit
Time Frame: Up to Month 6
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Emergency Departments (EDs)
Arm/Group | Control | PRIM-ER
Number analyzed (Participants) | 50458 | 48464
Number analyzed (Emergency Departments (EDs)) | 33 | 3
Proportion of participants | 0.281 | 0.287

7. Secondary Outcome: Survival: Time-to-event
Description: Number of days from index ED visit to death among those who died within six months following the index ED visit (Count of days)
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Emergency Departments (EDs)
Arm/Group | Control | PRIM-ER
Number analyzed (Participants) | 50458 | 48464
Number analyzed (Emergency Departments (EDs)) | 33 | 33
Days | 17.3 (38.8) | 17.1 (37.7)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse event (serious and non-serious) information data were not collected among participants in this retrospective study.
Arm/Group | Control | PRIM-ER
All-Cause Mortality (participants affected / at risk) | 14179/50458 | 13910/48464
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03424109/Prot_SAP_000.pdf